CLINICAL TRIAL: NCT04843072
Title: Balloon Expandable vs. Self Expanding Transcatheter Valve for Degenerated Bioprosthesis. THE BASELINE TRIAL.
Brief Title: Balloon vs. Self Expanding Transcatheter Valve for Degenerated Bioprosthesis
Acronym: BASELINE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Nicolas van Mieghem, Prof. dr., Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BASELINE TRIAL
Record Dates: First submitted 2021-03-24; First posted 2021-04-13 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Valve Heart Disease
MeSH Terms: conditions — Heart Valve Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Evolut R/Pro bioprosthesis (Experimental): Study subjects will receive a self-expanding-valve (either the Evolut R or PRO device)
  Interventions: Device: Evolut R/PRO bioprosthesis
- Edwards Sapien S3/Ultra bioprosthesis (Active Comparator): Study subjects will receive a balloon-expanding-valve (either the Edwards Sapien S3 or Ultra)
  Interventions: Device: Edwards Sapien S3/Ultra bioprosthesis

INTERVENTIONS:
Device: Evolut R/PRO bioprosthesis — To compare Evolut R/PRO versus Sapien S3/Ultra in failing surgical bioprostheses
  Arms: Evolut R/Pro bioprosthesis
Device: Edwards Sapien S3/Ultra bioprosthesis — Edwards Sapien S3/Ultra bioprosthesis
  Arms: Edwards Sapien S3/Ultra bioprosthesis

SUMMARY:
Transcatheter aortic valve implantation (TAVI) serves a growing spectrum of patients with symptomatic severe aortic stenosis (AS). Approximately 80% of surgical aortic valve replacements is performed using a bioprosthesis1. Durability of surgical bioprostheses varies based on the patient's age at the moment of implantation, type and size etc2. TAVI has become the preferred treatment for degenerated aortic bioprostheses in elderly patients3. The median time since index surgical aortic valve replacement (SAVR) and for bioprosthetic valve degeneration is typically 8 - 10 years4-6. TAVI in this setting has proven to have equally favorable results as in native aortic valves7. Balloon expandable8 and self-expanding9 transcatheter heart valves (THV) can be used in a degenerated bioprosthesis and each have specific assets and limitations. TAVI in a failed bioprosthesis can cause coronary obstruction, THV migration, paravalvular leakage and prosthesis patient mismatch. The SAPIEN-3 / Ultra and EVOLUT R/Pro are the 2 most commonly used THV platforms in contemporary clinical practice including treatment of failing surgical aortic bioprostheses.

Objective: To compare TAVI with EVOLUT R/Pro vs. SAPIEN-3 / Ultra in terms of device success.

Study design: International multi-center randomized study with 1:1 randomization to TAVI with SAPIEN-3 / Ultra or Evolut R/Pro.

Study population: 440 patients with a failing surgical aortic bioprosthesis (aortic stenosis with or without aortic regurgitation) and selected for transfemoral TAVI by heart-team consensus.

Investigational intervention: Transfemoral TAVI with SAPIEN-3 / Ultra or Evolut R/PRO

Main study parameters/endpoints:

1. Primary endpoint is device success at 30 days

   Defined by
   * Absence of procedural mortality AND
   * Correct positioning of a single prosthetic heart valve into the proper anatomical location AND
   * Intended performance of the prosthetic heart valve (no severe prosthesis- patient mismatch and mean aortic valve gradient < 20 mmHg or peak velocity < 3 m/s, AND no moderate or severe prosthetic valve regurgitation). Severe prosthesis patient mismatch is defined by effective orifice area (EOAi) ≤0.65 cm2/m2
2. Safety endpoint at 1 year defined by the composite of all-cause death, disabling stroke, rehospitalization for heart failure or valve related problems.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years
* Failing surgical aortic bioprosthesis requiring valve replacement and eligible for transfemoral TAVI with balloon expandable or self-expanding platform per heart team consensus based on multi-modality imaging assessment (including echocardiography and multidetector CT).
* Written informed consent

Exclusion Criteria:

* Not eligible for Transfemoral TAVI with SAPIEN-3 / Ultra and Evolut R/Pro
* Multi-valve defects requiring intervention
* Clinically unstable and/or inotropic/vasopressor /mechanical support.
* Known mural thrombus in the left ventricle
* Presence of a mechanical aortic valve
* History of recent (within 1 month) stroke or TIA

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Device success | 30 days post transcatheter valve implantation
  Device success, definition modified from VARC-2 criteria:
  * Absence of procedural mortality AND
  * Correct positioning of a single prosthetic heart valve into the proper anatomical location AND
  * Intended performance of the prosthetic heart valve (no severe prosthesis- patient mismatch and mean aortic valve gradient < 20 mmHg or peak velocity < 3 m/s, AND no moderate or severe prosthetic valve regurgitation). Severe prosthesis patient mismatch is defined by effective orifice area (EOAi) ≤0.65 cm2/m2

SECONDARY OUTCOMES:
Composite of all-cause death, disabling stroke, rehospitalization for heart failure or valve related problems | 1 year post transcatheter valve implantation
  Safety endpoint

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Van Mieghem, MD, PhD, Principal Investigator — Erasmus Medical Centre; Rutger-Jan Nuis, MD, PhD, Principal Investigator — Erasmus Medical Centre
Locations (14):
- Cedars Sinai, Los Angeles, California, United States
- Vienna General Hospital, Vienna, Austria
- St Paul's and Vancouver General Hospital, Vancouver, Canada
- Rigshospitalet, Copenhagen, Denmark
- Institut Cœur Poumon, Lille, France
- Germany (2):
  - Division of Cardiology, Pulmonology, and Vascular Medicine, Heinrich Heine University Medical Center Dusseldorf, Dusseldorf, Germany, Düsseldorf
  - University Hospital Mainz, Mainz
- Department of Cardiology, Onassis Cardiac Surgery Center, Athens, Greece, Athens, Greece
- Italy (2):
  - Interventional Cardiology Unit, Cardiovascular Department, Fondazione Poliambulanza Institute, Brescia, Italy, Brescia
  - University Hospital of Padova, Padua
- Erasmus Medical Centre, Rotterdam, Netherlands
- Centro Hospitalar de Lisboa Ocidental, Lisbon, Portugal
- Inselspital, University Hospital, Bern, Switzerland
- Leeds Teaching Hospitals, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nuis RJ, van Belle E, Teles R, Blackman D, Veulemans V, Santos IA, Pilgrim T, Tarantini G, Saia F, Iakovou I, Mascherbauer J, Vincent F, Geleijnse M, Sathananthan J, Wood D, Makkar R, Van Mieghem NM; BASELINE Investigators. BAlloon expandable vs. SElf expanding transcatheter vaLve for degenerated bioprosthesIs: design and rationale of the BASELINE trial. Am Heart J. 2023 Feb;256:139-147. doi: 10.1016/j.ahj.2022.11.013. Epub 2022 Nov 19. PMID 36410441